CLINICAL TRIAL: NCT05517538
Title: COMPARISON BETWEEN THE EFFICACY AND DURATION OF COSMETIC BOTULINUM TOXIN TYPE A INJECTION WITH AND WITHOUT ELECTROMYOGRAPHIC GUIDANCE
Brief Title: Split-face Study: Cosmetic Botulinum Toxin Type A Injection Under Electromyography-guidance Versus Conventional Palpation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Hayder Oleish Salih (Other)
Responsible Party: Sponsor-Investigator, Mohamed Hayder Oleish Salih, Masters Student, Alexandria University
Organization: Alexandria University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0106811
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Glabellar Frown Lines; Rhytides; Wrinkle; Facial Expression
Keywords: Botulinum Toxin; EMG-Guided Botulimun toxin injection; Cosmetic Botulinum toxin; Glabellar Merz Scale
MeSH Terms: conditions — Facial Expression | interventions — Botulinum Toxins, Type A; Botulinum Toxins; incobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: Split-Face: comparing two neurotoxin injection techniques, conventional palpation vs. EMG-guided injection.
  Follow up using EMG analysis and Glabellar Merz Scales
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palpation-guided (Experimental): injected with the Palpation Method of neurotoxin adminstration
  Interventions: Drug: Botulinum toxin type A
- EMG-guided (Experimental): injected with the EMG-guided Method of neurotoxin adminstration
  Interventions: Device: Electromyography-Needle Intramuscular Drug guidance; Drug: Botulinum toxin type A

INTERVENTIONS:
Device: Electromyography-Needle Intramuscular Drug guidance — EMG-guided needle neurotoxin injection
  Other Names: Electromyography-guided injection
  Arms: EMG-guided
Drug: Botulinum toxin type A — Botulinum toxin type A injection into the Corrugator Supercilii muscle
  Other Names: Botulinum neurotoxin; BoNT - A; BTX - A

SUMMARY:
The aim of this study was to compare between the conventional palpation method of botulinum toxin type A injection and the electromyography-guided method using clinical parameters and electromyography analysis.

DETAILED DESCRIPTION:
The study was conducted on 15 healthy-looking female subjects with visible glabellar rhytids when frowning. All participants were recruited from the outpatient clinic of Dermatology Department, Main University Hospital, Faculty of Medicine, Alexandria University. The mean age was 46.27 ± 6.31 with a range from 33 to 59 years. All 15 subjects completed the study.

Each subject provided a right and left corrugator supercilii muscles to the study. Each muscle was divided into a body and a tail, each part injected separately (n=60).

Neurotoxin injection into the corrugator body and tail by palpation method on one side and under EMG-guidance on the other.

Photographs were taken both at rest, and while frowning at each visit: pre-operatively, after 2 weeks and after 3 months.

Clinical grading according to static and dynamic Merz glabellar frown line scales and EMG analysis was done at each visit: pre-operatively, after 2 weeks and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Consent.
* Patients within age range of 25 - 60 years.
* Visible corrugator muscle rhytids when frowning by examination.

Exclusion Criteria:

* Patients with no, or minimal wrinkles on the studied area.
* Previous use of botulinum toxin in the previous 6 months.
* Patients on regular or very occasional antispasmodics.
* Patients with any neuromuscular disorders, infections or skin problems at the injection site.
* Patients with any known neurological disease.
* Patients who undergone surgery involving the glabellar area.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Interferance pattern Envelop amplitude (IPEA) | 3 months
  difference between + and - spikes in the EMG waveform [microvolt]
Muscle activity percentage (MAp) | 3 months
  percentage difference between the IPEA at follow up and base line [%]

SECONDARY OUTCOMES:
Glabellar Merz scales | 3 months
  Glabellar Merz scales : Dunamic and static [0-4]

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Oleish, MB BCh, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No